CLINICAL TRIAL: NCT06269770
Title: Multimodal Analgesia in TKA. The Role of Tapentadol
Brief Title: Tapentadol vs Tramadol in Total Knee Arthroplasty
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of Thessaly (Other)
Responsible Party: Principal Investigator, Elena Arnaoutoglou, Professor in Anesthesiology, University of Thessaly
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Tapentadol
Record Dates: First submitted 2024-02-03; First posted 2024-02-21 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Total Knee Replacement; Post-operative Pain; Chronic Pain
Keywords: total knee replacement; post-operative pain; tramadol; tapentadol
MeSH Terms: conditions — Pain, Postoperative; Chronic Pain | interventions — Tapentadol; Tramadol

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tramadol (Active Comparator): Tramadol will be administered in a multimodal analgesic approach to manage postoperative pain.
  Interventions: Drug: Tramadol
- Tapentadol (Active Comparator): Tapentadol will be administered in a multimodal analgesic approach to manage postoperative pain.
  Interventions: Drug: Tapentadol

INTERVENTIONS:
Drug: Tapentadol — Add tapentadol, for effective pain management in a multimodal setting during TKR.
  Arms: Tapentadol
Drug: Tramadol — Add tramadol, for effective pain management in a multimodal setting during TKR.
  Arms: Tramadol

SUMMARY:
Compare the effectiveness of tapentadol and tramadol as part of a multimodal analgesia treatment for Total Knee Replacement (TKR).

DETAILED DESCRIPTION:
As the population ages and becomes more active, the demand for TKR surgery is expected to increase. However, the treatment of TKR pain remains a challenge.

Postoperative pain is associated with longer hospital stays, lower satisfaction, increased opioid consumption, and transition to chronic pain. In TKR, the risk of chronic pain can be as high as 20%.

A suggested method of anesthesia and pain relief is the use of spinal anesthesia along with multimodal analgesia that includes an adductor canal block.

In our hospital, the multimodal analgesia protocol consists of intraoperative sedation with dexmedetomidine, a low dose of ketamine, paracetamol, NSAIDs, and magnesium. Dexamethasone and droperidol are preferred as antiemetics as they can improve the analgesic outcome.

To minimize the use of opioids, the administration of tramadol used to be the standard of care. Tapentadol is an opioid that can be equally effective in the treatment of postoperative pain and reduces the incidence of chronic pain after TKR.

ELIGIBILITY:
Inclusion Criteria:

* Patients for elective TKR
* ASA PS I - III

Exclusion Criteria:

* Patient refusal
* Cognitive disfunction
* Severe psychiatric disease
* Under medication with MAO inhibitors, tricyclic antidepressants, serotonin reuptake inhibitors
* Not speaking Greek
* Known allergy to the study drugs
* Contraindications for any of the study drugs
* Chronic renal failure (GFR < 50 ml/h)
* Liver failure
* Known regular use or misuse of opioids
* Pregnant women
* Patients undergoing general anesthesia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Post-operative pain | 6 hours after surgery
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 12 hours after surgery
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 1st postoperative day
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 2nd postoperative day
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 3rd postoperative day
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)

SECONDARY OUTCOMES:
Post-operative pain | 3 weeks after surgery
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 6 weeks after surgery
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Post-operative pain | 6 months after surgery
  Visual Analogue Scale (VAS) score measures 0 to 10 (0=no pain, 10=the worst pain)
Neuropathic pain | 6 months after surgery
  PainDETECT (0-35)
Quality of life postoperatively | 6 months after surgery
  Patient Quality 15 (0-150)
Patient Satisfaction | 5 days after surgery at Discharge
  5-point Likert scale (0-5) [5 representing higher satisfaction]
Depression | 5 days after surgery at Discharge
  Patient Health Questionnaire 9 (PHQ9) (0-27) [The higher the score, more severe the depression]
Function | 6 weeks after surgery
  Oxford Knee Score (OKS) (0-48)
Outcome | 6 weeks after surgery
  Knee Injury and Osteoarthritis Outcome Score (KOOS) (0-100)
Arthritis impact | 6 weeks after surgery
  ARTHRITIS IMPACT MEASUREMENT SCALES 2 Short Form (AIMS2-SF) (5Likert scale
Health Status | 6 weeks after surgery
  5 level EuroQol 5 Dimensions 5 level Score (EQ-5D-5L) (0-100) [The higher the score, the worse the health status]
Pain severity | 6 weeks after surgery
  Western Ontario and McMaster Universities Osteoarthritis (WOMAC) (0-96) [The higher the score the higher the disability due to osteoarthritis]

CONTACTS AND LOCATIONS:
Overall Officials: Eleni Arnaoutolglou, MD, PhD, Study Chair — Department of Anesthesiology, Faculty of Medicine, School of Health Sciences, University of Thessaly; Metaxia Bareka, MD, PhD, Principal Investigator — Department of Anesthesiology, Faculty of Medicine, School of Health Sciences, University of Thessaly
Locations (1):
- University Hospital Of Larissa, Larissa, Thessaly, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Baratta JL, Gandhi K, Viscusi ER. Perioperative pain management for total knee arthroplasty. J Surg Orthop Adv. 2014 Spring;23(1):22-36. doi: 10.3113/jsoa.2014.0022. PMID 24641894
- [Background] Roulet L, Rollason V, Desmeules J, Piguet V. Tapentadol Versus Tramadol: A Narrative and Comparative Review of Their Pharmacological, Efficacy and Safety Profiles in Adult Patients. Drugs. 2021 Jul;81(11):1257-1272. doi: 10.1007/s40265-021-01515-z. Epub 2021 Jul 1. PMID 34196947
- [Background] Rian T, Skogvoll E, Hofstad J, Hovik L, Winther SB, Husby VS, Klaksvik J, Egeberg T, Sand K, Klepstad P, Wik TS. Tapentadol vs oxycodone for postoperative pain treatment the first 7 days after total knee arthroplasty: a randomized clinical trial. Pain. 2021 Feb 1;162(2):396-404. doi: 10.1097/j.pain.0000000000002026. PMID 32773594